CLINICAL TRIAL: NCT07372469
Title: The Effect of Psychodrama on Mental Health Promotion in Nursing Students: A Randomized Controlled Trial
Brief Title: Psychodrama for Mental Health Promotion in Nursing Students
Acronym: PD-NURS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, ÖZGE KARACA, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PD-NURS-2024-01
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Promotion
Keywords: Psychodrama; Nursing students; Mental health; Psychosocial intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment and data analysis were conducted by an independent researcher who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychodrama Group (Experimental): Participants in this group received a structured psychodrama-based group intervention conducted once weekly for 12 weeks. The program was organized around thematic sessions including communication skills, self-awareness, self-esteem, personal development, values, family and close relationships, peer relationships, stress coping, anger management, assertiveness, sexuality, and physical well-being. Sessions involved experiential psychodramatic techniques such as role-playing, group games, and guided enactments aimed at enhancing emotional expression, interpersonal awareness, coping skills, and mental health promotion.
  Interventions: Behavioral: Psychodrama Group
- Presentation Group (Active Comparator): Participants in this group participated in weekly group sessions conducted concurrently with the intervention group for 12 weeks. Students prepared and delivered group presentations on topics aligned with the themes addressed in the psychodrama sessions. Presentations were shared in a classroom setting and followed by moderated group discussions. No psychodrama techniques, role-playing, or dramatic enactments were used.
  Interventions: Behavioral: Presentation Group

INTERVENTIONS:
Behavioral: Psychodrama Group — A psychodrama-based group intervention delivered in weekly sessions, using experiential techniques such as role-playing and guided enactments to support mental health promotion.
  Arms: Psychodrama Group
Behavioral: Presentation Group — Participants received a group-based educational intervention delivered once weekly for 12 weeks. Students prepared group presentations based on themes related to mental health promotion, which were presented in a classroom setting and followed by moderated group discussions. Psychodrama techniques, role-playing, or dramatic enactments were not used.
  Arms: Presentation Group

SUMMARY:
This randomized controlled trial aimed to examine the effect of a psychodrama group intervention on mental health promotion among nursing students. Participants were randomly assigned to an intervention group or a control group. The intervention group received weekly psychodrama sessions for 12 weeks, while the control group prepared group presentations on the same themes without psychodrama techniques. Mental health promotion levels were assessed before and after the intervention using a validated scale.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial conducted among nursing students. Participants were randomly assigned to either an intervention group or a control group. The intervention group participated in a psychodrama group intervention consisting of 12 weekly sessions, each lasting approximately 120-150 minutes. Sessions were facilitated by a trained psychodramatist and followed the classical psychodrama structure, including warm-up, action, and sharing phases.

The control group participated in weekly group presentations and discussions on the same themes as the intervention group but did not receive any psychodrama techniques. Mental health promotion levels were assessed before and after the intervention using the validated Mental Health Promotion Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student
* Aged 18 years or older
* Voluntary participation in the study

Exclusion Criteria:

* Being under 18 years of age
* Not being a nursing student

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Mental Health Promotion Level | Baseline and immediately after the 12-week intervention
  Mental health promotion levels were assessed before and after the intervention using the Mental Health Promotion Scale, a validated self-report instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Çağlar Şimşek, PhD, Principal Investigator — Istanbul Provincial Directorate of Health
Locations (1):
- Istanbul Kent University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No